CLINICAL TRIAL: NCT00397852
Title: Treatment of Stable Dislocated Both-Bone Distal Forearm Fractures in Children: A Randomized Trial Between Treatment With en Without Kirschner-Wires
Brief Title: Dislocated Stable Distal Both-Bone Forearm Fractures in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colaris, Joost, M.D. (Individual)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: colaris05
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2006-11-10 (Estimated); Status verified 2006-11

CONDITIONS: Fracture; Forearm; Distal; Child; Treatment
Keywords: Fracture; Forearm; Distal; Child; Treatment
MeSH Terms: conditions — Fractures, Bone | interventions — Bone Wires; Nuclear Receptor Subfamily 4, Group A, Member 2

INTERVENTIONS:
Procedure: Kirschner-wires or not

SUMMARY:
We create a randomized clinical trial between treatment with and without Kirschner wire fixation of a stable dislocated distal both-bone forearm fracture.

DETAILED DESCRIPTION:
children who arrive at the emergency unit with a dislocated both-bone distal forearm fracture will be asked to join the trial.

After informed consent, a randomization between 2 kinds of treatment will be done: K-wire fixation or no K-wire fixation of the fracture after a stable reposition.

Outpatient clinic visits till a follow-up of 6 months. During these visits we will investigate: the number of re-dislocations, re-operations, consolidation and dislocation on X-ray, function of both arms, complains in daily living and complications.

ELIGIBILITY:
Inclusion Criteria:

* both-bone forearm fracture
* distal
* dislocated
* stable after reposition
* age < 16 years

Exclusion Criteria:

* fracture older than 1 week
* no informed consent
* refracture
* open fracture (Gustillo 2 and 3)
* both fractures of type torus

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110
Dates: Start 2006-01

PRIMARY OUTCOMES:
re-operations/ re-dislocations

SECONDARY OUTCOMES:
pronation and supination
complications, function, esthetics, complains in daily living, X-rays

CONTACTS AND LOCATIONS:
Overall Officials: joost w colaris, drs, Principal Investigator
Locations (2):
- Netherlands (2):
  - Erasmus Medical Centre location Sophia Children's hospital, Rotterdam, South Holland
  - HAGA, location Juliana Children's Hospital, The Hague, South Holland